CLINICAL TRIAL: NCT01320878
Title: A Randomized Controlled Study of Inhaled Iloprost for the Treatment of Pulmonary Hypertension After Repair of Congenital Heart Disease
Brief Title: Study of Inhaled Iloprost for the Treatment of Pulmonary Hypertension After Repair of Congenital Heart Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xu Zhuoming, Director of Cardiac intensive Care Unit,Department of Thoracic and Cardiovascular Sugery,Shanghai Children's Medical Center., Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SJTUMS-10-16
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Iloprost

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- iloprost low dose group (Active Comparator): iloprost 30 ng/kg/min inhalation for 10 minutes,q4h in day time and q6h at night for 2 days
  Interventions: Drug: iloprost nebuliser solution
- iloprost high dose group (Active Comparator): iloprost 50 ng/kg/min inhalation for 10 minutes, q4h in day time and q6h at night for 2 days
  Interventions: Drug: iloprost nebuliser solution
- placebo group (Placebo Comparator): distilled water 2 ml per session
  Interventions: Drug: distilled water

INTERVENTIONS:
Drug: iloprost nebuliser solution — iloprost 30 ng/kg/min inhalation for 10 minutes,q4h in day time and q6h at night for 2 days
  Other Names: Ventavis
  Arms: iloprost low dose group
Drug: iloprost nebuliser solution — iloprost 50 ng/kg/min inhalation for 10 minutes, q4h in day time and q6h at night for 2 days
  Other Names: Ventavis
  Arms: iloprost high dose group
Drug: distilled water — distilled water 2 ml per session
  Other Names: Treeful
  Arms: placebo group

SUMMARY:
The objective of this study was to assess the efficacy and appropriate dose of iloprost for inhalation in the treatment of postoperative pulmonary hypertension in children with congenital heart defects.

DETAILED DESCRIPTION:
Pulmonary hypertension is a serious postoperative complication in children with congenital heart defects, which has a high incidence and mortality. Iloprost is a prostacyclin analogue. When applied by inhalation, it selectively dilates pulmonary vessels, without side affecting the systemic circulation. No randomized controlled trials (RCT) of iloprost have previously been performed in this indication. The investigators study is the first RCT of iloprost for inhalation after surgery of children's congenital heart diseases to be performed in this field.

ELIGIBILITY:
Inclusion Criteria:

Before corrective procedure for CHD, two of bellow ten criteria should be met:

* Decreased respiratory infection & decreased exercise tolerance
* Pulse SaO2 < 93% in left-right shunt CHD case (in room air)
* EKG: right ventricular hypertrophy, right atrial dilatation
* Chest X-ray: enhanced vascular signs in trans-hilar, loss of blood vessel in bilateral lung fields, pulmonary arterial trunk dilatation, right ventricular enlargement
* Cardiac echocardiography: fast tricuspid or pulmonary valve regurgitant velocity, ventricular and aortic level bidirectional shunt, or even right-to-left shunt
* Underfilling of pulmonary capillary, 'pruning' of the peripheral blood vessels
* Pp/Ps > 0.75
* Qp/Qs <1.5
* PVR > 9WU/m2
* Rp/Rs > 0.5

Exclusion Criteria:

* a body weight of < 2 kg,
* prematurity (birth 36 weeks postconceptual age)
* renal dysfunction (creatinine >= 1.5 mg/dL 48 hours before surgery)
* PLT < 50,000*109/L and obvious bleeding
* LCOS or hypotension on arrival to the intensive care unit

After corrective procedure for CHD:

* deficient anatomy associated with remained intracardiac shunts and severe artrio-ventricular regurgitation
* severe arrhythmia led to low cardiac output

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2007-10; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
all cause pulmonary artery pressure | one year

SECONDARY OUTCOMES:
central venous pressure | one year
blood pressure | one year
cardiac index | one year
pulmonary vascular resistance | one year
mortality | one year

CONTACTS AND LOCATIONS:
Overall Officials: Zhuo-ming Xu, MD,PhD, Study Director — Cardiac intensive Care Unit,Department of Thoracic and Cardiovascular Sugery,Shanghai Children's Medical Center
Locations (1):
- Cardiac intensive Care Unit,Department of Thoracic and Cardiovascular Sugery,Shanghai Children's Medical Center, Shanghai, China

REFERENCES:
- [Result] Gorenflo M, Gu H, Xu Z. Peri-operative pulmonary hypertension in paediatric patients: current strategies in children with congenital heart disease. Cardiology. 2010;116(1):10-7. doi: 10.1159/000313864. Epub 2010 Apr 24. PMID 20424447